CLINICAL TRIAL: NCT04601428
Title: CSR02-Fab-TF as Hepatic Intra-arterial Therapy in Intermediate Stage B or Limited Advanced Stage C Hepatocellular Carcinoma (HCC): Dose-Escalation Study to Assess Safety and Tolerability
Brief Title: Hepatic IA Therapy in Stage B or Limited Stage C Hepatoma (HCC)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Koo Foundation Sun Yat-Sen Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF-CSR02-001
Record Dates: First submitted 2020-09-29; First posted 2020-10-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular carcinoma; HCC; hepatoma; IA (intra-arterial) therapy; PLVAP; CSR02-Fab-TF
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: The dose escalation phase of the study will begin with 3 single cohort subjects and then proceed to a traditional 3 +3 study design until a Maximum Tolerated Dose (MTD) or an active dose (i.e., a dose at which subjects achieve a complete response in the liver or complete elimination of tumor blood flow) is identified. Once an appropriate dose in established, an expansion phase will administer CSR02-Fab-TF to 16 additional subjects to estimate the response proportion in subjects with refractory HCC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Arm (Experimental)
  Interventions: Biological: IA therapy of HCC with CSR02-Fab-TF

INTERVENTIONS:
Biological: IA therapy of HCC with CSR02-Fab-TF — Intra-Arterial Infusion of CSR02-Fab-TF

SUMMARY:
Intra-arterial (IA) therapy is generally used to treat HCC tumors that are too extensive to excise or treat with potentially curative local therapy. IA therapy takes advantage of the fact that the blood supply of HCC comes predominantly from the hepatic artery compared with the surrounding normal liver which is predominantly supplied by portal venous blood. The intent is to deprive the HCC of its blood supply, leading to the death of the tumor. Traditionally, various methods have been used to block the HCC blood supply, but improvements are needed. This study will investigate a new agent designed in the laboratory to block only tumor blood vessels, not blood vessels in the normal liver.

DETAILED DESCRIPTION:
Genetic testing was done to identify differences between HCC tumors and normal liver, and a protein, PLVAP, was shown to be present on the blood vessels of HCC but not on the blood vessels of normal liver. An antibody, CSR02, was made that recognizes PLVAP and then the Fab portion of that antibody was combined with tissue factor, a normal human protein that initiates the clotting cascade. The result is a manufactured (recombinant) protein called CSR02-Fab-TF. Preclinical studies in a mouse model showed that infusion of an equivalent mouse protein resulted in the necrosis (death) of a transplanted human HCC. The current study is designed first, to identify a safe and optimal dose of CSR02-Fab-TF in patients , and then second, to determine the response rate of HCC tumors to the IA administration of CSR02-Fab-TF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of HCC by at least one of the following criteria:

  * Histological confirmation;
  * Magnetic resonance imaging (MRI) or computerized tomography (CT) consistent with liver cirrhosis AND at least one solid liver lesion > 1 cm with intense contrast uptake during the arterial phase followed by contrast washout during the venous phase regardless of alpha-fetal protein (AFP) level
* Barcelona Clinic Liver Cancer (BCLC) Intermediate Stage B or limited Advanced Stage C (see Protocol Section 3.1). Patients with Stage C disease should have received or been offered and chosen not to receive systemic therapy
* Inadequate response to prior liver-directed therapy (e.g., TACE, bland embolization, Y90, ablation, radiation therapy) to the same targeted area or progressive disease after prior liver-directed therapy) or to one or more systemic therapies
* Not a candidate for curative resection, liver transplantation, or percutaneous ablation (See Protocol Appendix 3)
* Eastern Collective Oncology Group (ECOG) performance status ≤1 (See Protocol Appendix 5)
* Adequate laboratory parameters, including:

  * Serum total bilirubin ≤ 2x ULN
  * Alkaline phosphatase, aspartate aminotransferase (AST) and aspartate aminotransferase (ALT) < 5 x ULN;
  * Serum creatinine ≤ 1.5 mg/dL;
  * Prothrombin time (international normalized ratio; INR) ≤ 1.5;
  * Absolute neutrophil count > 1000/μL;
  * Platelet count > 75,000/μL;
  * Hgb > 8 g/dL
* Acceptable pulmonary status, including room air O2 saturation > 90%
* Child-Pugh A-B7 without clinically significant ascites (See Protocol Appendix 4)
* Signed informed consent
* All subjects must be surgically sterile, at least two years post-menopausal (if female), or agree to use adequate, effective contraception approved by the Investigator until two (2) months after receiving a final dose of CSR02-Fab-TF

Exclusion Criteria:

* Eligible for transplantation by Milan criteria (Protocol Appendix 3) or potentially eligible if successfully "down staged" by pre-transplant therapy
* Prior organ transplantation
* Any small molecule drug treatment for HCC (including TACE) within the previous 30 days, treatment with biological agents or any investigational therapy within the previous 60 days, or treatment with Y90 within the previous 90 days.
* Previously treated malignancies from which the subject has not been disease-free for at least 2 years, except for adequately treated non-melanoma skin cancer, in situ cancer, or low-grade prostate or bladder cancer
* Severe chronic obstructive or other pulmonary disease with hypoxemia that requires supplementary oxygen or clinically significant pleural effusions
* New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 3 months prior to therapy, unstable arrhythmia, symptomatic peripheral arterial vascular disease, or presence of an artificial or other vascular device requiring chronic anticoagulation (See Protocol Appendix 6)
* Any of the following risks related to QT/QTc interval:

  * Baseline prolongation of QT/QTc interval (repeated interval > 480 milliseconds using Frederica's QT correction formula);
  * History of additional risk factors for Torsades de Pointes (e.g. heart failure, hypokalemia, family history of Long QT syndrome);
  * Concomitant medications that have a known risk for prolongation of the QT/QTc interval (see https://crediblemeds.org/new-drug-list/)
* Major surgery, vascular injury, or serious illness within the previous 60 days
* Known inherited thrombophilia (hypercoagulable state) or history of unprovoked venous or arterial thrombosis
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy at screening. Subjects with prior HBV (positive HBSAg) must have HBV viral load < 2000 IU/mL or be receiving concurrent anti-HBV therapy to be eligible. Subjects on anti-HBV therapy must have been on treatment with a viral load maintained at < 2000 IU/mL for at least 4 weeks prior to first dose and continue on this same therapy throughout study treatment. Subjects with HCV infection are eligible if other eligibility criteria are met
* Females who are breast-feeding
* Allergy to iodinated contrast medium that is uncontrolled or refractory to medical therapy
* Therapeutic anticoagulation that cannot be stopped 24-72 hours before treatment (per Section 4.5) and reinstituted no sooner than 72 hours after therapy
* Any concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events from intra-arterial infusion of CSR02-Fab-TF in patients with hepatoma only or largely confined to the liver, and resistant/recurrent after prior therapy | Infusion to Day 50
  Measured by the number of treatment-emergent adverse events and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
HCC blood flow | MRI on Day 4
  HCC blood flow will be assessed by magnetic resonance imaging (MRI) on day 4 after infusion of CSR02-FabTF.

SECONDARY OUTCOMES:
Determine tumor response to intra-arterial infusion of CSR02-Fab-TF | by MRI on Day 50 and then every 3 months for an average of one year.
  Measured by radiographic response using acceptable imaging modalities used for assessment of tumor vasculature and blood flow (MRI or CT) based on mRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Weiden, M.D., Study Director — KFSYSCC consultant
Locations (4):
- Taiwan (4):
  - National Cheng Kung University Hospital (NCKUH), Tainan, North Dist.
  - Koo Foundation Sun Yat-Sen Cancer Center (KFSYSCC), Taipei, Pei-Tou Dist.
  - National Taiwan University Hospital (NTUH), Taipei, Zhongzheng Dist.
  - KFSYSCC, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forner A, Gilabert M, Bruix J, Raoul JL. Treatment of intermediate-stage hepatocellular carcinoma. Nat Rev Clin Oncol. 2014 Sep;11(9):525-35. doi: 10.1038/nrclinonc.2014.122. Epub 2014 Aug 5. PMID 25091611
- [Background] Wang YH, Cheng TY, Chen TY, Chang KM, Chuang VP, Kao KJ. Plasmalemmal Vesicle Associated Protein (PLVAP) as a therapeutic target for treatment of hepatocellular carcinoma. BMC Cancer. 2014 Nov 6;14:815. doi: 10.1186/1471-2407-14-815. PMID 25376302
- See also: PubMed ID: 25091611 Treatment of intermediate-stage hepatocellular carcinoma — https://doi.org/10.1038/nrclinonc.2014.122
- See also: PubMed ID: 25376302 Plasmalemmal Vesicle Associated Protein (PLVAP) as a therapeutic target for treatment of hepatocellular carcinoma — https://doi.org/10.1186/1471-2407-14-815